CLINICAL TRIAL: NCT02155322
Title: A Phase II Study of Pegylated Interferon Alfa-2b in AJCC Stage III (TxN1-2M0) Melanoma Subjects After Regional Lymph Node Dissection in Russia
Brief Title: A Phase II Study of Pegylated Interferon Alfa-2b for the Adjuvant Treatment of Melanoma Subjects in Russia (MK-4031-400)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4031-400
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-IFN (Experimental): 6.0 μg/kg/week subcutaneous administration during the Induction Phase of 8 weeks followed by a dose of 3.0 μg/kg/week subcutaneous administration in the Maintenance Period (Week 8 to Month 12)
  Interventions: Biological: Pegylated Interferon Alfa-2b

INTERVENTIONS:
Biological: Pegylated Interferon Alfa-2b — 6 μg/kg, weekly dosing, subcutaneous administration, Induction Phase - first 8 weeks
Biological: Pegylated Interferon Alfa-2b — 3 μg/kg SC once weekly for a 42-week maintenance phase (for a total treatment of up to approximately 1 year)

SUMMARY:
This study will assess the safety of Pegylated Interferon Alfa-2b (PEG-IFN) as an adjuvant treatment for melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Competent to self-administer the subcutaneous injections of PEG-IFN
* Histologically documented involved regional lymph nodes of a primary cutaneous melanoma or unknown primary, meeting the study's staging criteria
* Had the primary melanoma completely resected with adequate surgical margins and undergone operation for positive regional lymph nodes within 84 days of study start
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1
* Adequate hepatic, renal and bone marrow function as defined by study parameters obtained within 4 weeks prior to study start
* For a female subject who is of childbearing potential or male participant with female sexual partner who is of childbearing potential, agree to use acceptable methods of contraception for at least 2 weeks prior to study start and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations

Exclusion Criteria:

* Mucous membrane melanoma or ocular melanoma
* Known hypersensitivity to the components of study drug (including acetaminophen), or its analogs
* Evidence of distant or non-regional lymph node metastases or in-transit metastases
* Disease that cannot be completely surgically resected
* Prior malignancy within the past 5 years other than surgically cured non-melanoma skin cancer or cervical carcinoma in situ
* Severe cardiovascular disease, i.e. arrhythmias, requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease
* Hepatic decompensation
* Thyroid dysfunction not responsive to therapy
* Uncontrolled diabetes mellitus
* Clinically active autoimmune disease
* Clinically active and/or uncontrolled infection, including active hepatitis
* Human immunodeficiency virus (HIV)
* History of neuropsychiatric disorder requiring hospitalization
* Actively abusing alcohol or drugs
* Pregnant, lactating, or of reproductive potential and not using an effective means of contraception
* Medical condition requiring chronic systemic corticosteroids
* Received any experimental therapy within 30 days prior to enrolling in this study
* Received any prior chemotherapy, immunotherapy, hormonal or radiation therapy for melanoma
* Previously received interferon-α for any reason
* Known serious hypersensitivity reaction to PEG-IFN or interferon alfa-2b

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled Russian participants with malignant melanoma who had undergone surgical resection and lymphadenectomy.
Groups:
- PEG-IFN: Participants received PEG-IFN 6 μg/kg subcutaneously (SC) once weekly during an 8-week induction phase followed by 3 μg/kg SC once weekly for a 42-week maintenance phase (treatment up to approximately 1 year).
Period: Overall Study
Arm/Group | PEG-IFN
Started | 33
Treated | 32 (32 of 33 participants treated. 1 participant not treated at the discretion of the investigator.)
Completed | 19
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Relapse/Recurrence | 8
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: An adverse event was any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: From first dose through follow-up; up to 13 months
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN
Number analyzed (Participants) | 32
Percentage of participants | 100.0

2. Primary Outcome: Percentage of Participants Discontinuing Study Drug Because of AEs
Description: as for outcome 1
Time Frame: From first dose to last dose of treatment; up to 12 months
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN
Number analyzed (Participants) | 32
Percentage of participants | 3.1

ADVERSE EVENTS:
Time Frame: From first dose through follow-up; up to 13 months
Description: AEs for all participants who received at least one dose of study drug.
Arm/Group | PEG-IFN
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN (N=32)
MONOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
LEUKOCYTURIA (Renal and urinary disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
LEUKOPENIA (Blood and lymphatic system disorders) | 9 (11)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (9)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (9)
NAUSEA (Gastrointestinal disorders) | 7 (8)
ASTHENIA (General disorders) | 12 (12)
FATIGUE (General disorders) | 7 (15)
INFLUENZA LIKE ILLNESS (General disorders) | 7 (42)
INJECTION SITE ERYTHEMA (General disorders) | 6 (8)
PYREXIA (General disorders) | 26 (62)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 17 (32)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 17 (34)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (3)
DIZZINESS (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 4 (6)
DEPRESSION (Psychiatric disorders) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.